CLINICAL TRIAL: NCT04755413
Title: Use of Biomarker Risk Score to Optimize Therapy in Patients With Coronary Artery Disease: The Precision CAD Trial
Brief Title: The Precision CAD Trial
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Arshed A. Quyyumi, Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: STUDY00001179
Record Dates: First submitted 2021-02-11; First posted 2021-02-16 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Biomarkers
MeSH Terms: conditions — Coronary Artery Disease | interventions — Behavior Therapy; Standard of Care; Registries

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Optimization Group (Experimental): Participants with CAD and a BRS greater than 0 who are randomized to the Optimization Group have treatment goals that include achieving LDL-C<70 mg/dL, hemoglobin A1c <7%, blood pressure <130/80 mmHg, smoking cessation, at least 30 minutes of moderate-intensity aerobic activity 5 days a week and weight loss to body mass index <30 kg/m2. To achieve these goals, both pharmacological and lifestyle interventions will be considered and individualized for each patient.
  Interventions: Other: Medical/Behavioral therapy
- Usual Care Group (Active Comparator): Participants with CAD and a BRS greater than 0 who are randomized to the usual care group will receive standard of care therapy prescribed by their primary care physician and/or cardiologist. Patients and their physicians will be informed that their BRS is ≥1 and they have been randomized to the usual care group.
  Interventions: Other: Standard of Care
- Registry Group (Other): Participants with BRS of 0 at baseline and after 3 months will undergo follow-up including measurements of BRS at the time-points specified for the randomized subjects and also for adverse events. Laboratory results and questionnaire data will be obtained on the phone.
  Interventions: Other: Registry

INTERVENTIONS:
Other: Medical/Behavioral therapy — * Sedentary lifestyle: Advise increasing exercise to at least 30 minutes of moderate-intensity aerobic activity 5 days a week.
  * Overweight/Obese: Advise calorie reduction, dietician consultation.
  * Smoking: standard smoking cessation advice and literature and medical therapy as indicated to include Wellbutrin, nicotine patch etc.
  * High LDL cholesterol: a) Start high dose statin if patient not on high dose statin.
    b) If on high dose statin, add ezetimibe 10mg daily c) If statin intolerant, start ezetimibe 10mg, colestid or other bile sequestrant combination.
    d) If still not at goal, start PCSK-9 inhibitor e) LDL cut off of <55mg/dl in diabetes
  * Blood Pressure optimization treatment following 2020 International Society of Hypertension Global Hypertension Practice Guidelines.
  * Diabetes management: HbA1c goal 6.5%
  Arms: Optimization Group
Other: Standard of Care — Participants will receive standard of care therapy prescribed by their primary care physician and/or cardiologist.
  Arms: Usual Care Group
Other: Registry — Participants with BRS of 0 will get measurements of BRS at the time-points specified for the randomized subjects and also for adverse events.
  Arms: Registry Group

SUMMARY:
People with Coronary Artery Disease (CAD) have narrow or blocked arteries that supply blood to the heart. Reduced blood flow to the heart muscle from CAD can cause chest pain or aching, especially with exercise or activity. CAD can lead to weakening of the heart muscle or heart failure, and a higher risk of heart attack or death. Certain proteins in the blood, known as biomarkers, can be found in people with CAD. Higher levels of these biomarkers are associated with a greater risk of complications from CAD. The purpose of this study is to see if a customized treatment based on biomarkers will reduce the biomarker levels and lead to lower risk of complications from CAD.

DETAILED DESCRIPTION:
People with Coronary Artery Disease (CAD) have narrow or blocked arteries that supply blood to the heart. Reduced blood flow to the heart muscle from CAD can cause chest pain or aching, especially with exercise or activity. CAD can lead to weakening of the heart muscle or heart failure, and a higher risk of heart attack or death. Certain proteins in the blood, known as biomarkers, can be found in people with CAD. Higher levels of these biomarkers are associated with a greater risk of complications from CAD. The purpose of this study is to see if a customized treatment based on biomarkers will reduce the biomarker levels and lead to lower risk of complications from CAD.

Participants with high biomarker levels will be randomly assigned (like flipping a coin) to either the treatment group or usual care. Both groups will have physical exams, blood tests, and answer questionnaires. Participants in the treatment group will have their medications adjusted based on their biomarker levels. They will also be asked to make lifestyle changes like diet, exercise, and quitting smoking. Participants in the usual care group will receive the standard of care prescribed by their doctor.

This study will take place in research rooms at Emory University Hospital and the Woodruff Memorial Research Building.

Participants will be paid for being in the study.

Participants will be recruited from Emory Healthcare outpatient cardiology clinics and cath labs. Participants will be identified through the medical record and by their doctors. Written consent will be obtained from Participants before they can join the study.

Study data and blood samples will be collected and banked for possible research in the future. These may also be shared with other researchers including researchers outside of Emory.

This study will advance scientific knowledge and benefit human health by giving us more treatment options for CAD.

ELIGIBILITY:
Inclusion Criteria:

* Individuals aged 21-90 years with stable CAD.
* Patients with any amount of atherosclerosis via coronary angiogram or coronary computed tomography angiography (CCTA).
* Patients undergoing revascularization therapy or recent acute coronary syndrome (ACS) will be eligible for recruitment and will be recruited at least 4 weeks after admission for an ACS or percutaneous intervention and 3 months after coronary bypass graft surgery.
* Patients with CAC levels ≥ 400

Exclusion Criteria:

* Planned revascularization,
* New York Heart Association class III or IV heart failure symptoms,
* LVEF <40%,
* eGFR<45,
* Pregnancy, congenital heart disease, severe symptomatic valvular heart disease, active malignancy and cardiac transplant.

Ages: 21 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 276 (Actual)
Dates: Start 2022-10-19 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Change in plasma levels of hsCRP | Baseline, 1 year post intervention
  Blood will be drawn for measurement of plasma levels of hsCRP to compare the optimization group and the usual care group.
Change in plasma levels of hs-cTnI | Baseline, 1 year post intervention
  Blood will be drawn for measurement of plasma levels of hs-cTnI to compare the optimization group and the usual care group.
Change in plasma levels of BNP | Baseline, 1 year post intervention
  Blood will be drawn for measurement of plasma levels of BNP to compare the optimization group and the usual care group.
Change in plasma levels of suPAR | Baseline, 1 year post intervention
  Blood will be drawn for measurement of plasma levels of suPAR to compare the optimization group and the usual care group.
Change in Biomarker Risk Score (BRS) | Baseline, 1 year post intervention
  The BRS score is a simple and manual observation of 4 biomarker results above a predetermined cutpoint that are run on FDA cleared and or CE marked platforms. The BRS is calculated using levels of the 4 biomarkers. Biomarker levels will be considered abnormal if hsCRP is >3 mg/L, suPAR (pg/mL) >2863 (males) and >4063 (women), hs-TnI (pg/mL)> 6.3 (men), >5.5 (women), and BNP (pg/mL) >122 (men), >184.1 (women). The BRS ranges from 0 to 4 based on the number of biomarkers that are elevated above these cut off values. Higher score correlates with worse outcome.
Change in composite complications | Baseline, 1,3,6,9 months post intervention and 1,2,3,5 years post intervention
  Difference in rates of composite of CV death/MI/ heart failure hospitalizations, stroke/ revascularization between optimization group, usual care group and registry group.

SECONDARY OUTCOMES:
Change in plasma levels of hsCRP | Baseline, 1, 3, 6, 9 months post intervention and 2, 3, 5 years post intervention
  Blood will be drawn for measurement of plasma levels of hsCRP to compare the optimization group and the usual care group.
Change in plasma levels of hs-cTnI | Baseline, 1, 3, 6, 9 months post intervention and 2, 3, 5 years post intervention
  Blood will be drawn for measurement of plasma levels of hs-cTnI to compare the optimization group and the usual care group.
Change in plasma levels of BNP | Baseline, 1, 3, 6, 9 months post intervention and 2, 3, 5 years post intervention
  Blood will be drawn for measurement of plasma levels of BNP to compare the optimization group and the usual care group.
Change in plasma levels of suPAR | Baseline, 1, 3, 6, 9 months post intervention and 2, 3, 5 years post intervention
  Blood will be drawn for measurement of plasma levels of suPAR to compare the optimization group and the usual care group.
All cause death | 5 years post intervention
  All cause death at 5 years in the optimization group compared to usual care group.

CONTACTS AND LOCATIONS:
Overall Officials: Arshed Quyyumi, MD, Principal Investigator — Emory University
Locations (5):
- United States (5):
  - Emory Johns Creek Hospiatl, Atlanta, Georgia
  - Emory University Hospital Midtown, Atlanta, Georgia
  - Emory University Hospital, Atlanta, Georgia
  - The Emory Clinic, Atlanta, Georgia
  - Emory Saint Joseph's Hospital, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No